CLINICAL TRIAL: NCT02464163
Title: Phase 1/2 Adaptive Design Trial to Evaluate the Immunogenicity and Safety of Panblok (H7 rHA) at Three Dose Levels Adjuvanted With a Stable Oil-in-Water Emulsion Compared With Unadjuvanted H7 rHA in Healthy Adults Aged 18 and Older
Brief Title: Trial to Evaluate the Immunogenicity and Safety of Panblok® (H7 rHA) in Healthy Adults Aged 18 and Older
Acronym: PSC26
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSC26
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Panblok 30µg in 2% SE (Experimental): 30µg recombinant hemagglutinin in a 2% oil-in-water stable emulsion (rHA adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: Panblok; Biological: rHA adjuvant
- Panblok 15µg in 2% SE (Experimental): 15µg recombinant hemagglutinin in a 2% oil-in-water stable emulsion (rHA adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: Panblok; Biological: rHA adjuvant
- Panblok 7.5µg in 2% SE (Experimental): 7.5µg recombinant hemagglutinin in a 2% oil-in-water stable emulsion (rHA adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: Panblok; Biological: rHA adjuvant
- Panblok 30µg (No Adjuvant) (Experimental): 30µg recombinant hemagglutinin (no adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: Panblok

INTERVENTIONS:
Biological: Panblok — Intramuscular injection
  Other Names: recombinant hemagglutinin; rHA
Biological: rHA adjuvant — Intramuscular injection
  Other Names: SE
  Arms: Panblok 15µg in 2% SE; Panblok 30µg in 2% SE; Panblok 7.5µg in 2% SE

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of a recombinant hemagglutinin (rHA) influenza vaccine derived from A/Anhui/1/2013 (H7N9) administered at 3 dose levels in adjuvanted (SE) rHA formulations and 1 dose levels in an unadjuvanted rHA formulation.

DETAILED DESCRIPTION:
All currently licensed influenza vaccines in the United States are produced in embryonated hen's eggs. There are several well-recognized disadvantages to the use of eggs as the substrate for influenza vaccine. Eggs require specialized manufacturing facilities and could be difficult to scale up rapidly in response to an emerging need such as a pandemic. It is usually necessary to adapt candidate vaccine viruses for high-yield growth in eggs, a process that can be time consuming, is not always successful, and can select receptor variants that may have suboptimal immunogenicity. In addition, agricultural diseases that affect chicken flocks, and that might be an important issue in a pandemic due to an avian influenza virus strain, could easily disrupt the supply of eggs for vaccine manufacturing. Therefore, development of alternative substrates for influenza vaccine production has been identified as a high-priority objective.

One potential alternative method for production of influenza vaccine is expression of the influenza virus hemagglutinin (HA) using recombinant DNA techniques. This alternative avoids dependence on eggs and is very efficient because of the high levels of protein expression under the control of the baculovirus polyhedrin promoter.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, regardless of gender, aged 18 years and above
2. Able to give written informed consent to participate.
3. Body temperature <100.0ºF.
4. The subject must be in reasonably good health as determined by targeted physical examination, when necessary, based on medical history.
5. Women of child-bearing potential (WOCBP) must have a negative urine pregnancy test within 24 hours preceding receipt of first and second vaccine doses.
6. Women are considered not of child-bearing potential if they are:

   * Surgically sterile
   * Menopausal, defined as no natural menses for ≥12 months
7. Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits and remote contacts.

Exclusion Criteria:

1. Persons who previously received an H5N1 or H7N9 influenza vaccine or who plan to receive an H5N1or H7N9 influenza vaccine while participating in the study.
2. Persons who plan to receive a seasonal influenza vaccine earlier than Day 42 of participation in this study, i.e. before the post-vaccination serology sample is obtained.
3. Persons with an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of immune responses.
4. Persons taking medications or treatments that may adversely affect the immune system, e.g. cytotoxic agents, immunosuppressive doses of corticosteroids, anti-TNFα agents.
5. Persons with an active neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years.
6. Persons with a history of documented autoimmune disease.
7. Women currently pregnant, nursing mothers or women planning a pregnancy between enrollment and 42 days after randomization.
8. Persons who have had a prior serious reaction to any influenza vaccine.
9. Persons with a known history of Guillain-Barré Syndrome (GBS).
10. Persons with a history of anaphylactic-type reaction to injected vaccines.
11. Persons with a history of illicit drug use or alcohol abuse that may compromise the subject's ability to comply with the protocol.
12. Persons who received a seasonal influenza vaccine < 6 months prior to enrollment (may delay enrollment).
13. Persons who received any licensed inactivated or recombinant (non-live) vaccine within 2 weeks prior to enrollment or any licensed live vaccine within 1 month prior to enrollment (may delay enrollment) (See separate exclusion criteria #1 and #12 for seasonal and H5N1 influenza vaccines.)
14. Persons who have had an acute illness or fever (>38º C or >100º F) within three days prior to study enrollment (enrollment may be delayed for full recovery, if acceptable to investigator).
15. Persons currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication) or have received an experimental agent within 1 month prior to enrollment in this study, or who expect to receive another experimental agent during participation, or intend to donate blood during the 42-day primary study period.
16. Persons who received immunoglobulin or another blood product within the 3 months prior to enrollment in this study. Persons who expect to receive immunoglobulin or another blood product during the 42-day primary period of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Treanor, MD, Principal Investigator — University of Rochester Center for Vaccine Studies
Locations (9):
- United States (9):
  - Coastal Clinical Research, Mobile, Alabama
  - Avail Clinical Research, DeLand, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Meridian Clinical Research, Omaha, Nebraska
  - Regional Clinical Research, Inc., Endwell, New York
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Benchmark Reseach, Austin, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panblok 30µg in 2% SE | Panblok 15µg in 2% SE | Panblok 7.5µg in 2% SE | Panblok 30µg (No Adjuvant)
Started | 102 | 102 | 102 | 101
Completed | 99 | 94 | 97 | 96
Not Completed | 3 | 8 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Modified Per Protocol Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Panblok 7.5µg in 2% SE | Panblok 15µg in 2% SE | Panblok 30µg in 2% SE | Panblok 30µg (No Adjuvant) | Total
Number analyzed (Participants) | 95 | 94 | 99 | 94 | 382
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: <65 Years | 45 | 45 | 49 | 42 | 181
  Age, Categorical: >=65 Years | 50 | 49 | 50 | 52 | 201
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 54 | 56 | 61 | 233
  Male | 33 | 40 | 43 | 33 | 149

OUTCOME MEASURES:

1. Primary Outcome: Demonstrate That the Immunogenicity of Adjuvanted Panblok H7 rHA is Sufficient to Support Emergency Use Authorization in the Event of a Declared Pandemic.
Description: The primary endpoint will be "seroprotection rate" to the selected dose of adjuvanted H7 rHA, defined by a post-vaccination HAI titer ≥40 on Day 42. The definition of success will be a lower bound of the two-sided 95% CI ≥ 70% for adults <65 and ≥60% for adults ≥65 years of age.
Time Frame: 42 Days
Population: Modified Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Panblok 7.5µg in 2% SE | Panblok 15µg in 2% SE | Panblok 30µg in 2% SE | Panblok 30µg (No Adjuvant)
Number analyzed (Participants) | 95 | 94 | 99 | 94
Participants | 11 | 9 | 15 | 1

2. Secondary Outcome: Reactogenicity Immediately After Each Injection, Extending to Day 7
Description: Solicited events of local and systemic reactogenicity Days 0-7
Time Frame: 7 Days
Population: Reactogenicity Population
Measure: Count of Participants; unit: Participants
Arm/Group | Panblok 7.5µg in 2% SE | Panblok 15µg in 2% SE | Panblok 30µg in 2% SE | Panblok 30µg (No Adjuvant)
Number analyzed (Participants) | 100 | 101 | 101 | 97
Participants
  7 Days After First Vaccination | 37 | 33 | 33 | 27
  7 Days After Second Vaccination | 30 | 30 | 26 | 18

3. Secondary Outcome: Long-term Safety Assessed by Incidence of SAEs, NOCIs. AESs Over 12 Months Following Vaccination
Time Frame: 13 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Panblok 7.5µg in 2% SE | Panblok 15µg in 2% SE | Panblok 30µg in 2% SE | Panblok 30µg (No Adjuvant)
Number analyzed (Participants) | 100 | 101 | 102 | 97
Participants
  Angina unstable | 0 | 0 | 1 | 0
  Myocardial infarction | 0 | 0 | 0 | 1
  Sinus bradycardia | 0 | 0 | 1 | 0
  Chest pain | 0 | 0 | 1 | 0
  Appendicitis | 1 | 0 | 0 | 0
  Cellulitis | 0 | 1 | 0 | 0
  Rib fracture | 1 | 0 | 0 | 0
  Upper limb fracture | 0 | 0 | 0 | 1
  Arthralgia | 1 | 0 | 0 | 0
  Fracture malunion | 0 | 1 | 0 | 0
  Musculoskeletal pain | 1 | 0 | 0 | 0
  Osteoarthritis | 2 | 0 | 0 | 0
  Osteolysis | 0 | 1 | 0 | 0
  Cervicobrachial syndrome | 1 | 0 | 0 | 0
  Syncope | 0 | 0 | 1 | 0
  VIIth nerve paralysis | 1 | 0 | 0 | 0
  Suicide attempt | 0 | 1 | 0 | 0
  Peripheral arterial occlusive disease | 0 | 0 | 1 | 0

4. Secondary Outcome: Unsolicited Adverse Events (UAEs) During Days 0-42 Following the First Administration of Study Vaccine
Description: Unsolicited adverse events (UAEs) Days 0-42.
Time Frame: 42 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Panblok 7.5µg in 2% SE | Panblok 15µg in 2% SE | Panblok 30µg in 2% SE | Panblok 30µg (No Adjuvant)
Number analyzed (Participants) | 100 | 101 | 102 | 97
Participants
  Cardiac disorders | 0 | 0 | 1 | 0
  Ear and labyrinth disorders | 1 | 0 | 0 | 0
  Endocrine disorders | 0 | 2 | 0 | 0
  Eye disorders | 0 | 0 | 1 | 0
  Gastrointestinal disorders | 5 | 2 | 2 | 4
  General disorders | 4 | 2 | 1 | 2
  Immune system disorders | 1 | 0 | 0 | 0
  Infections and infestations | 6 | 6 | 4 | 0
  Injury, poisoning and procedural complications | 3 | 3 | 2 | 0
  Investigations | 0 | 2 | 0 | 0
  Metabolism and nutrition disorders | 1 | 1 | 0 | 0
  Musculoskeletal and connective tissue disorders | 4 | 2 | 5 | 1
  Neoplasms benign, malignant and unspecified | 1 | 2 | 0 | 0
  Nervous system disorders | 3 | 2 | 5 | 1
  Psychiatric disorders | 0 | 0 | 0 | 1
  Reproductive system and breast disorders | 0 | 1 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 6 | 2 | 1 | 1
  Skin and subcutaneous tissue disorders | 1 | 0 | 2 | 1
  Vascular disorders | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 0 to Week 55
Arm/Group | Panblok 7.5µg in 2% SE | Panblok 15µg in 2% SE | Panblok 30µg in 2% SE | Panblok 30µg (No Adjuvant)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/101 | 0/102 | 1/97
Serious Adverse Events (participants affected / at risk) | 4/100 | 4/101 | 3/102 | 2/97
Other Adverse Events (participants affected / at risk) | 0/100 | 0/101 | 0/102 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panblok 7.5µg in 2% SE (N=100) | Panblok 15µg in 2% SE (N=101) | Panblok 30µg in 2% SE (N=102) | Panblok 30µg (No Adjuvant) (N=97)
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No